CLINICAL TRIAL: NCT05495464
Title: A Pilot "Window-3" Study of Acalabrutinib Plus Rituximab Followed by Brexucabtagene Autoleucel Therapy in Patients With Previously Untreated High-risk Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Kite, A Gilead Company (Industry); Acerta Pharma, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0872; NCI-2022-06281 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-07-28; First posted 2022-08-10 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma; Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — acalabrutinib; Rituximab; brexucabtagene autoleucel; Cyclophosphamide; fludarabine phosphate; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acalabrutinib and Rituximab (Part 1) (Experimental): Participants may receive acalabrutinib and rituximab for up to 12 cycles. Each cycle is 28 days.
  Interventions: Drug: Acalabrutinib; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate
- Brexucabtagene Autoleucel (Part 2) (Experimental): Participants will have a procedure called leukapheresis to collect enough T cells.
  Interventions: Other: Brexucabtagene Autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate

INTERVENTIONS:
Drug: Acalabrutinib — Given by PO
  Arms: Acalabrutinib and Rituximab (Part 1)
Drug: Rituximab — Given by IV (vein)
  Other Names: Rituxan
  Arms: Acalabrutinib and Rituximab (Part 1)
Other: Brexucabtagene Autoleucel — Given by IV (vein)
  Arms: Brexucabtagene Autoleucel (Part 2)
Drug: Cyclophosphamide — Given by IV (vein)
  Other Names: Cytoxan®; Neosar®
Drug: Fludarabine Phosphate — Given by IV (vein)
  Other Names: Fludarabine; Fludara®

SUMMARY:
To learn if giving acalabrutinib, rituximab, and brexucabtagene autoleucel to patients with previously untreated high-risk mantle cell lymphoma (MCL) can help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To determine the safety profile of the acalabrutinib plus rituximab combination followed by CAR T-cell therapy in newly diagnosed high risk MCL patients.

SECONDARY OBJECTIVES:

To evaluate efficacy measured by complete response (CR) rate and progression free survival (PFS) of the acalabrutinib plus rituximab combination followed by CAR T-cell therapy in newly diagnosed high risk MCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of mantle cell lymphoma by hematopathology. MCL should have CD20 positivity (by flow or IHC in tissue or in BM) with presence of chromosome translocation t(11;14), (q13;q32) and/or overexpression of cyclin D1 in tissue biopsy (See Appendix I, footnote 10).
2. Newly diagnosed high risk patient without any prior therapy for MCL and are eligible to receive AR and CART cell therapy.
3. High risk MCL (Blastoid/pleomorphic histology, high Ki-67 (≥50%), TP53/NOTCH1/2, NSD2, UBR5, FAT1, TRAF2, SP140, POT1, SMARCA4, KMT2D, BIRC3 mutated or any of these mutations or more than 2 mutations with some evidence of prognostic impact, complex karyotype and/or Bulky disease >= 5 cm, FISH positive for TP53 or MYC from involved tissues or TP53 and MYC positive intensity in lymphoma cells in involved tissues (positive by hem-path criteria at MDACC), high risk MIPI score (with Ki-67%). Presence of any or all of these features would qualify as high risk but will need to be reviewed and approved by the study PI. (We will not use any assay which is not FDA approved or not CLIA certified to determine the eligibility of these patients)
4. Patients who are eligible to receive CAR T therapy
5. Patients who are willing and able to participate in all required evaluations and procedures in this study protocol, including swallowing capsules and tablets without difficulty.
6. Understand and voluntarily sign an IRB-approved informed consent form.
7. Age ≥ 18 years at the time of signing the informed consent.
8. Bi-dimensional measurable disease using the 2014 Cheson criteria (Measurable disease by PET-CT scan defined as at least 1 lesion that measures ≥ 1.5 cm in single dimension.) Spleen only involved (>=20 cm), these patients are allowed if they meet other high-risk features, determined by the study PI.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 1 or less (See Appendix IV).
10. An absolute neutrophil count (ANC) > 1,000/mm3 and platelet count >100,000/mm3 (Patients who have >50% bone marrow or spleen infiltration by MCL are eligible if their ANC is ≥ 500/mm3 [growth factor allowed] or their platelet level is equal to or >= than 30,000/mm3. These patients should be discussed with the PI of the study for final approval).
11. Serum bilirubin <1.5 mg/dl and Cr Clearance ≥ 60 mL/min by Cockroft-Gault Formula (Appendix VIII) or by >=60 ml/min by 24 hour urine Cr clearance test (Appendix VIII) , AST (SGOT) and ALT (SGPT) < 2.5 x upper limit of normal or < 5 x upper limit of normal if hepatic metastases are present. Gilbert's disease is allowed.
12. Women of childbearing potential (WOBP) must have a negative serum or urine pregnancy test. WOBP and males must be willing to use highly effective methods of birth control. Woman of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and for 2 days after the last dose of acalabrutinib and for 12 months following the last dose of rituximab and 6 months after the completion of CAR T infusion. For male patients with a pregnant or non-pregnant WOCBP partner, should use barrier contraception, during treatment and for 2 days after the last dose of acalabrutinib and for 1 month following the last dose of rituximab and 6 months after the completion of CAR T infusion even if they have had a successful vasectomy. (see Appendix VII).
13. Cardiology cleared for receiving acalabrutinib and CART

EXCLUSION CRITERIA PART 1:

1. Isolated bone marrow or GI only disease MCL patients and/or lack of measurable disease.
2. Pregnant or breast-feeding females.
3. Patients who are primary refractory to AR (No response/progressive disease within first 4 months of AR)
4. Received any investigational drug within 30 days or 5 half-lives (whichever is shorter) before first dose of study drug.
5. Current life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the subject's safety or put the study at risk.
6. Known HIV infection.
7. Patients who do not meet high risk features as indicated above. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HBsAg) negative will need to have a negative polymerase chain reaction (PCR) and must be willing to undergo DNA PCR testing during the study to be eligible. Those who are HBsAg positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result to be eligible. Those who are hepatitis C PCR positive will be excluded.
8. Prior malignancy (or any other malignancy requiring active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ ca prostate, in situ melanoma (> 5 mm margins) or other cancer from which the subject has been disease free for ≥ 3 years or which will not limit survival to < 3 years.
9. Central nervous system involvement with mantle cell lymphoma or with suspected or confirmed progressive multifocal leukoencephalopathy (PML). Magnetic resonance imaging (MRI) of the brain, if performed, showing evidence of central nervous system (CNS) lymphoma or Lumbar puncture with flow cytometry, if performed, with CSF involvement.
10. History or presence of CNS disorder, such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, cerebral edema, posterior reversible encephalopathy syndrome, or any autoimmune disease with CNS involvement.
11. Active bleeding, history of bleeding diathesis (such as Hemophilia or Von-Willebrand disease), Any history of intracranial bleed or stroke within 6 months of first dose of study drug.
12. Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura).
13. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction, or any other gastrointestinal condition that could interfere with the absorption and metabolism of acalabrutinib.
14. Presence of a clinically significant gastrointestinal ulcer diagnosed by endoscopy within 3 months before first dose of study drug.
15. Requires anticoagulation with warfarin or equivalent vitamin K antagonist, active treatment for pulmonary embolism (PE)/ deep vein thrombosis (DVT) and persons with mechanical cardiac valves.
16. History of symptomatic deep vein thrombosis (DVT) or pulmonary embolism requiring systemic anticoagulation within the last 6 months of enrollment
17. Concomitant use of corticosteroids at > 20 mg prednisone or equivalent per day longer than 2 weeks.
18. Primary immunodeficiency
19. History of confirmed autoimmune disease (e.g. Crohn's disease, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years. Rheumatology clearance required for pts with remote history of auto-immune disease.
20. History of severe, immediate hypersensitivity reaction attributed to aminoglycosides
21. The use of strong CYP3A inhibitors within 1 week or strong CYP3A inducers within 3 weeks of the first dose of study drug is prohibited.
22. Requires treatment with strong CYP3A inhibitors or inducers (refer to list in Appendix VI).
23. Any of the following cardiac related conditions:

    * NYHA Class III and IV heart failure (Appendix IX),
    * Active/symptomatic coronary artery disease,
    * Myocardial infarction in the preceding 6 months,
    * Significant conduction abnormalities, including but not limited to:

      * Left bundle branch block,
      * 2nd degree AV block type II,
      * 3rd degree block,
      * QT prolongation (QTc > 500 msec),
      * Sick sinus syndrome,
      * Ventricular tachycardia,
      * Symptomatic bradycardia (heart rate < 50 bpm),
      * Persistent and uncontrolled atrial fibrillation.
    * Uncontrolled hypertension
    * Uncontrolled Hypotension
    * Light headedness and syncope,
24. Acute infection requiring systemic anti-infective treatment systemic antibiotics, antivirals, or antifungals, or including subjects with positive cytomegalovirus [CMV] DNA polymerase chain reaction [PCR] within 14 days prior to initiation of therapy. Patient who exhibit active uncontrolled infection on AR alone will not be excluded but would await adequate infection control and then get CAR T, as long as they have evidence of disease.
25. Vaccinated with live, attenuated vaccines within 6 weeks of first dose of study drug.
26. Any other serious medical condition including, but not limited to, uncontrolled diabetes mellitus, COPD, renal failure, psychiatric illness or social circumstances that, in the investigator's opinion places the patient at unacceptable risk and would prevent the patient from signing the informed consent form or complying with study procedures.
27. Known history of hypersensitivity or anaphylaxis to study drug(s) including active product or excipient components.
28. Prothrombin time (PT)/INR or aPTT (in the absence of lupus anticoagulant) >2x ULN.
29. Concurrent participation in another therapeutic clinical trial.
30. Has difficulty with or is unable to swallow oral medication or has significant gastrointestinal disease that would limit absorption of oral medication.
31. Known history of hypersensitivity or anaphylaxis to study drug(s) including active product or excipient components.
32. Major surgical procedure within 28 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Within 30 days after CAR T-cell infusion
  Unacceptable toxicity is defined as any grade 3 or higher treatment related toxicities happened within 30 days after CAR T-cell infusion. Will monitor the unacceptable toxicity for two patient cohorts together using the Bayesian stopping boundaries calculated based on beta-binomial distribution. The regimen will be considered excessively toxic if the unacceptable toxicity rate at 30 days after CAR T infusion is above 30%. Frequency tables will be used to summarize categorical variables such as toxicity type/severity.

CONTACTS AND LOCATIONS:
Overall Officials: Preetesh Jain, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org